CLINICAL TRIAL: NCT02210156
Title: Effects of a Dietary Supplement on the Incidence of Acute Respiratory Infections in Susceptible Adults
Brief Title: Effects of a Supplement on Acute Respiratory Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omnilife Manufactura, SA de CV (Industry)
Collaborators: University of Guadalajara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Omnilife 01; 19/UG-JAL/2012 (Other: Registro Estatal de Investigacion. Secretaria de Salud. Gobierno de Jalisco. Mexico.)
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Respiratory Tract Infection
Keywords: Respiratory tract infection; Incidence; Dietary supplements; Micronutrients; Plant extracts
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Dietary Supplements; Micronutrients; Plant Extracts

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Two envelopes of the product in 240 ml of water in a disposable cup, 90 days of actual consumption.
  Interventions: Other: Placebo
- Omniplus Supreme (Experimental): Two envelopes of the product in 240 ml of water in a disposable cup, 90 days of actual consumption.
  Interventions: Dietary Supplement: Omniplus Supreme

INTERVENTIONS:
Dietary Supplement: Omniplus Supreme — Two dietitians prepared the products (one preparer per product) by dissolving two envelopes of 20 ml of the product in 240 ml of water in a disposable cup, every day from Monday to Saturday during the intervention period (90 days of actual consumption). In order to maintain blinding, these dietitians then gave the prepared cups to two different supervisors who in turn gave the product to each participant for consumption (once-daily doses). The preparation and delivery of the product was carried out during two work shifts (morning and afternoon), depending on each participants work schedule. The supervisors recorded product administration and consumption for each participant on a control form.
  Other Names: Food supplement with micronutrients and plant extracts
  Arms: Omniplus Supreme
Other: Placebo — A product with maltodextrins, flavors and colorants without vitamins, minerals and plant extracts. Two dietitians prepared the products (one preparer per product) by dissolving two envelopes of 20 ml of the product in 240 ml of water in a disposable cup, every day from Monday to Saturday during the intervention period (90 days of actual consumption). In order to maintain blinding, these dietitians then gave the prepared cups to two different supervisors who in turn gave the product to each participant for consumption (once-daily doses). The preparation and delivery of the product was carried out during two work shifts (morning and afternoon), depending on each participants work schedule. The supervisors recorded product administration and consumption for each participant on a control form.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the consumption of a nutritional supplement with micronutrients and herbal extracts has an effect on the incidence of acute respiratory infections in susceptible adults.

Our hypothesis is that subjects who consume the nutritional supplement will have a lower incidence and duration of acute respiratory infections in comparison with the placebo group.

DETAILED DESCRIPTION:
We conducted a randomized, parallel, double-blind, placebo-controlled, 90-day clinical trial from January to April, 2012. All staff who worked at the Omnilife's Entrepreneur Support Department (CREO by its initials in Spanish) were invited to participate. This department within Omnilife has a high incidence of acute respiratory infections (ARI) as reported internally by the company's medical service (accounting for 55% of doctor visits within the department in 2010) and hence, they represent a high number of individuals susceptible to ARI.

We held a preliminary session with the department's entire staff to explain the procedures; we asked subjects interested to participate in the study to sign an informed consent form and fill a clinical history. The latter included an assessment of stress, using the Perceived Stress Scale (in which higher scores indicate higher levels of stress), and physical activity, using the International Physical Activity Questionnaire or IPAQ (in which physical activity is categorized in three levels: light, moderate and vigorous).

In a second session the same week, participants visited the company's medical service for measurements of their weight and height (in accordance with the International Society for the Advancement of Kinanthropometry or ISAK standards), control laboratory tests and a medical examination to rule out the presence of infections. Weight measurements were taken using a Tanita BC553 Ironman Inner Scan Body Fat Scale (capacity of 150 kg, accuracy to 0.1 kg). Height measurements were made using a Seca 206 Stadiometer (accuracy to 0.1 cm, measuring range to 220 cm). Both measurements were performed by a two certified and standardized anthropometrists. Body mass index (BMI) was subsequently calculated using both variables as follows: BMI = weight in kg/(height in m)2.

The medical examination was performed by the attending physician and a nurse. It consisted of an assessment of vital signs following procedures described in the literature and a physical examination of bodily organs and systems. Temperature was measured using a Microlife MT 1931 digital thermometer (measuring range from 32 to 43.9°C, accuracy to 0.1°C). Heart and respiratory rates were measured using a 3M Littmann Classic II S.E. stethoscope. Blood pressure readings were taken using a 3M Littmann Classic II S.E. stethoscope and an Aneroid Sphygmomanometer ce0483 (18-300 mmHg measurement range, accuracy to 2 mmHg).

Laboratory tests were conducted with the support of an external laboratory (Instituto Diagnostico Especializado Arboledas, IDEA by its initials in Spanish). Included were a blood test of six items (fasting glucose, uric acid, creatinine, blood urea nitrogen, cholesterol and triglycerides) analyzed by the spectrophotometric method, a complete blood count with a flow cytometry/microscopy analysis of platelets, and a spectroscopy analysis to assess liver function. Subjects of laboratory analyses were tested after a 12-hour fast. This laboratory has obtained quality control certification from the Quality Assurance for Laboratories Program (PACAL) and the Internal Evaluation Quality Program (PREVECAL). In addition, its staff is certified in clinical diagnosis by the National Association of Clinical Chemists (CONAQUIC).

Subjects who met inclusion criteria were randomly assigned to two groups: one which received the supplement (n=30), and a control group who received a placebo, which consisted in a mixture of maltodextrins, colors and flavors. Every day two dietitians prepared the products, who then gave the prepared products to two different supervisors who in turn gave the product to each participant for consumption. The supervisors recorded product administration and consumption for each participant on a control form.

Simultaneously, each week the supervisors provided each participant with an ARI symptom and side effect diary to be filled in daily (indicating whether or not the symptom in question had presented). Participants delivered the supervisors their filled-in diaries the following week. Subjects were also requested not to self-medicate in the event they should feel any of the symptoms and to notify the principal researcher and attending physician, who would make a clinical assessment to confirm the presence or absence of ARI and provide any needed medical treatment. In such cases, participants were not to be excluded from the study, but treatment provided to them was documented. At the end of the supplementation period, the initial assessments were performed again. Subjects were also asked about their perceptions of their own health at that time compared to how they felt at the beginning of the study.

Quantitative variables are expressed as mean (SD). Qualitative variables are expressed as frequency (%). Fisher's exact test was used to compare distribution percentages of qualitative variables between groups and to compare the total proportion of ill subjects across intervention groups using intent-to-treat and per-population concepts. The risk ratio and the risk difference were also calculated for episodes of ARI. To compare the average of quantitative variables between treatments, the Mann-Whitney U test was used. Statistical analyzes were run using the SPSS program version 10 for Windows and Open Epi version 3.01; p<0.05 was considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects (without active respiratory infections, or without diseases that compromise immune system)
* Who presented no abnormalities in their laboratory tests (active infections, immunosuppression, renal or hepatic impairment)
* Who did not take drugs that affect the immune system (anti-inflammatory drugs, antibiotics, steroids).

Exclusion Criteria:

* Subjects with active acute respiratory infections.
* Subjects with chronic respiratory disease requiring treatment other than bronchodilators at the time of assessment.
* Subjects with diseases affecting the immune system (autoimmune illness, diabetes, etc.)
* Pregnant women or currently nursing.
* Subjects with cardiovascular disorders (uncontrolled hypertension) or neurological disorders (epilepsy).
* Subjects with allergies to any components of the products.
* Subjects with low treatment adherence (less than 80%).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Incidence of acute respiratory infections | 90 days
  Number of subjects with at least one episode of acute respiratory infection according to supplementation group.

SECONDARY OUTCOMES:
Mean episodes of acute respiratory infections | 90 days
  Mean episodes of acute respiratory infections by supplementation group
Mean duration of acute respiratory infections | 90 days
  Mean duration in days of acute respiratory infections by supplementation group
Number of subjects with more than one acute respiratory infection episode | 90 days
  Number of subjects with more than one acute respiratory infection episode by supplementation group
Absenteeism | 90 days
  Number of subjects who reported absenteeism because of acute respiratory infections, by supplementation group
Episode-related medication | 90 days
  Number of subjects who reported episode-related medication by supplementation group
Fasting glucose | 90 days
  Changes in fasting glucose (final vs initial)
Uric acid | 90 days
  Changes in uric acid (final vs initial)
Blood urea nitrogen | 90 days
  Changes in blood urea nitrogen (final vs initial)
Creatinine | 90 days
  Changes in creatinine (final vs initial)
Cholesterol | 90 days
  Changes in cholesterol (final vs initial)
Triglycerides | 90 days
  Changes in triglycerides (final vs initial)
Number of acute respiratory infections | 90 days
  Number of acute respiratory infections episodes by supplementation group.

CONTACTS AND LOCATIONS:
Overall Officials: María F. Bernal-Orozco, Ph.D., Study Director — Omnilife Manufactura, SA de CV; Margarita Posada-Falomir, B.Sc.(Nutr.), Principal Investigator — Omnilife Manufactura, SA de CV; Rafael Ortega-Orozco, M.D., Principal Investigator — Omnilife Manufactura, SA de CV; Elvia Silva-Villanueva, M.Sc.(O.H)., Principal Investigator — Omnilife Manufactura, SA de CV; Gabriela Macedo-Ojeda, Ph.D., Principal Investigator — University of Guadalajara; Yolanda F. Marquez-Sandoval, Ph.D., Principal Investigator — University of Guadalajara; Barbara Vizmanos-Lamotte, M.D., Ph.D, Principal Investigator — University of Guadalajara
Locations (1):
- Omnilife, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Eccles R. Understanding the symptoms of the common cold and influenza. Lancet Infect Dis. 2005 Nov;5(11):718-25. doi: 10.1016/S1473-3099(05)70270-X. PMID 16253889
- [Background] Calder PC, Kew S. The immune system: a target for functional foods? Br J Nutr. 2002 Nov;88 Suppl 2:S165-77. doi: 10.1079/BJN2002682. PMID 12495459
- [Background] Manoharan A, Winter J. Tackling upper respiratory tract infections. Practitioner. 2010 Nov;254(1734):25-8, 2-3. PMID 21166296
- [Background] Wintergerst ES, Maggini S, Hornig DH. Contribution of selected vitamins and trace elements to immune function. Ann Nutr Metab. 2007;51(4):301-23. doi: 10.1159/000107673. Epub 2007 Aug 28. PMID 17726308
- [Background] Ramirez MT, Hernandez RL. Factor structure of the Perceived Stress Scale (PSS) in a sample from Mexico. Span J Psychol. 2007 May;10(1):199-206. doi: 10.1017/s1138741600006466. PMID 17549893
- [Background] Stephen AI, Avenell A. A systematic review of multivitamin and multimineral supplementation for infection. J Hum Nutr Diet. 2006 Jun;19(3):179-90. doi: 10.1111/j.1365-277X.2006.00694.x. PMID 16756533
- [Background] Goyal SK, Samsher, Goyal RK. Stevia (Stevia rebaudiana) a bio-sweetener: a review. Int J Food Sci Nutr. 2010 Feb;61(1):1-10. doi: 10.3109/09637480903193049. PMID 19961353
- [Background] Gohil KJ, Patel JA, Gajjar AK. Pharmacological Review on Centella asiatica: A Potential Herbal Cure-all. Indian J Pharm Sci. 2010 Sep;72(5):546-56. doi: 10.4103/0250-474X.78519. PMID 21694984
- [Background] Cumashi A, Ushakova NA, Preobrazhenskaya ME, D'Incecco A, Piccoli A, Totani L, Tinari N, Morozevich GE, Berman AE, Bilan MI, Usov AI, Ustyuzhanina NE, Grachev AA, Sanderson CJ, Kelly M, Rabinovich GA, Iacobelli S, Nifantiev NE; Consorzio Interuniversitario Nazionale per la Bio-Oncologia, Italy. A comparative study of the anti-inflammatory, anticoagulant, antiangiogenic, and antiadhesive activities of nine different fucoidans from brown seaweeds. Glycobiology. 2007 May;17(5):541-52. doi: 10.1093/glycob/cwm014. Epub 2007 Feb 12. PMID 17296677
- [Background] Panossian A, Wikman G. Evidence-based efficacy of adaptogens in fatigue, and molecular mechanisms related to their stress-protective activity. Curr Clin Pharmacol. 2009 Sep;4(3):198-219. doi: 10.2174/157488409789375311. Epub 2009 Sep 1. PMID 19500070
- [Background] Karkos PD, Leong SC, Arya AK, Papouliakos SM, Apostolidou MT, Issing WJ. 'Complementary ENT': a systematic review of commonly used supplements. J Laryngol Otol. 2007 Aug;121(8):779-82. doi: 10.1017/S002221510600449X. Epub 2006 Nov 24. PMID 17125579
- [Background] Barrett B, Brown R, Rakel D, Mundt M, Bone K, Barlow S, Ewers T. Echinacea for treating the common cold: a randomized trial. Ann Intern Med. 2010 Dec 21;153(12):769-77. doi: 10.7326/0003-4819-153-12-201012210-00003. PMID 21173411
- [Background] Chandra RK. Nutrition and the immune system: an introduction. Am J Clin Nutr. 1997 Aug;66(2):460S-463S. doi: 10.1093/ajcn/66.2.460S. PMID 9250133
- [Background] Field CJ, Johnson IR, Schley PD. Nutrients and their role in host resistance to infection. J Leukoc Biol. 2002 Jan;71(1):16-32. PMID 11781377
- [Background] Rosler D, Fuchs N, Markolin G, Edler B, Kuklinski B, Kastenbauer T. [Reduction of influenza-like infections by a phytoextract-vitamin-combination: a randomized, double-blind, placebo-controlled study]. MMW Fortschr Med. 2012 Dec 17;154 Suppl 4:115-22. German. PMID 23326930
- [Background] Liu Y, Jing H, Wang J, Zhang R, Zhang Y, Zhang Y, Xu Q, Yu X, Xue C. Micronutrients decrease incidence of common infections in type 2 diabetic outpatients. Asia Pac J Clin Nutr. 2011;20(3):375-82. PMID 21859655
- [Background] Linday LA, Dolitsky JN, Shindledecker RD. Nutritional supplements as adjunctive therapy for children with chronic/recurrent sinusitis: pilot research. Int J Pediatr Otorhinolaryngol. 2004 Jun;68(6):785-93. doi: 10.1016/j.ijporl.2004.01.009. PMID 15126020
- [Background] Linday LA, Shindledecker RD, Tapia-Mendoza J, Dolitsky JN. Effect of daily cod liver oil and a multivitamin-mineral supplement with selenium on upper respiratory tract pediatric visits by young, inner-city, Latino children: randomized pediatric sites. Ann Otol Rhinol Laryngol. 2004 Nov;113(11):891-901. doi: 10.1177/000348940411301108. PMID 15562899
- [Background] Penny ME, Marin RM, Duran A, Peerson JM, Lanata CF, Lonnerdal B, Black RE, Brown KH. Randomized controlled trial of the effect of daily supplementation with zinc or multiple micronutrients on the morbidity, growth, and micronutrient status of young Peruvian children. Am J Clin Nutr. 2004 Mar;79(3):457-65. doi: 10.1093/ajcn/79.3.457. PMID 14985222
- [Background] Begin F, Santizo MC, Peerson JM, Torun B, Brown KH. Effects of bovine serum concentrate, with or without supplemental micronutrients, on the growth, morbidity, and micronutrient status of young children in a low-income, peri-urban Guatemalan community. Eur J Clin Nutr. 2008 Jan;62(1):39-50. doi: 10.1038/sj.ejcn.1602682. Epub 2007 Feb 14. PMID 17299460
- [Background] Graat JM, Schouten EG, Kok FJ. Effect of daily vitamin E and multivitamin-mineral supplementation on acute respiratory tract infections in elderly persons: a randomized controlled trial. JAMA. 2002 Aug 14;288(6):715-21. doi: 10.1001/jama.288.6.715. PMID 12169075
- [Background] Avenell A, Campbell MK, Cook JA, Hannaford PC, Kilonzo MM, McNeill G, Milne AC, Ramsay CR, Seymour DG, Stephen AI, Vale LD. Effect of multivitamin and multimineral supplements on morbidity from infections in older people (MAVIS trial): pragmatic, randomised, double blind, placebo controlled trial. BMJ. 2005 Aug 6;331(7512):324-9. doi: 10.1136/bmj.331.7512.324. PMID 16081445
- [Background] Croci DO, Cumashi A, Ushakova NA, Preobrazhenskaya ME, Piccoli A, Totani L, Ustyuzhanina NE, Bilan MI, Usov AI, Grachev AA, Morozevich GE, Berman AE, Sanderson CJ, Kelly M, Di Gregorio P, Rossi C, Tinari N, Iacobelli S, Rabinovich GA, Nifantiev NE; Consorzio Interuniversitario Nazionale per la Bio-Oncologia (CINBO), Italy. Fucans, but not fucomannoglucuronans, determine the biological activities of sulfated polysaccharides from Laminaria saccharina brown seaweed. PLoS One. 2011 Feb 28;6(2):e17283. doi: 10.1371/journal.pone.0017283. PMID 21387013
- [Background] Erickson KL, Medina EA, Hubbard NE. Micronutrients and innate immunity. J Infect Dis. 2000 Sep;182 Suppl 1:S5-10. doi: 10.1086/315922. PMID 10944478
- [Background] Lofgren E, Fefferman NH, Naumov YN, Gorski J, Naumova EN. Influenza seasonality: underlying causes and modeling theories. J Virol. 2007 Jun;81(11):5429-36. doi: 10.1128/JVI.01680-06. Epub 2006 Dec 20. No abstract available. PMID 17182688
- [Background] Nahas R, Balla A. Complementary and alternative medicine for prevention and treatment of the common cold. Can Fam Physician. 2011 Jan;57(1):31-6. PMID 21322286
- [Background] Puertollano MA, Puertollano E, de Cienfuegos GA, de Pablo MA. Dietary antioxidants: immunity and host defense. Curr Top Med Chem. 2011;11(14):1752-66. doi: 10.2174/156802611796235107. PMID 21506934
- [Background] Gestal-Otero JJ, Takkouche B, Blasco-Huelva P. Infecciones respiratorias agudas. Gripe. En: Piédrola-Gil G, editor. 1oa ed. Medicina preventiva y salud pública. Barcelona: Masson; 2001. p. 491-505
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] International Physical Activity Questionnaire [Web site]; 2005 [access november 4th 2011]. IPAQ Research Committee. Guidelines for data processing and analysis of the International Physical Activity Questionnaire (IPAQ). Short and long forms. Available in: http://www.ipaq.ki.se/scoring.pdf.
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Marfell-Jomes M, Olds T, Stewart A, Carter L. Estándares internacionales para la evaluación antropométrica. Revisión 2008. South Africa: Sociedad Internacional para el Avance de la Cineantropometría; 2008.
- [Background] World Health Organization [Web site]. Geneva: The Organization; 2006 [updated november 11th 2011; access november 11th 2011]. BMI classification. Available in: http://apps.who.int/bmi/index.jsp?introPage=intro_3.html.
- [Background] Vizmanos B, Bernal MF. Signos vitales. In: López-Uriarte P, Hunot C, Altamirano M, Macedo G, Vizmanos B, editors. Manual de prácticas de evaluación del estado nutricio. 1st ed. Guadalajara: La noche; 2007. p. 25-30.
- [Background] Gupta S, Rajauria G, Sbu-Ghannam N. Study of the microbial diversity and antimicrobial properties of Irish edible brown seaweeds. Int J Food Sci Technol. 2010;45:482-9.
- [Background] Jensen GS, Ginsberg DJ, Huerta P, Citton M, Drapeau C. Consumption of Aphanizomenon flos-aquae has rapid effects on the circulation and function of immune cells in humans. A novel approach to nutritional mobilization of the immune system. JANA 2000;2:50-8.
- [Background] Castelloti C. Algas. Su uso terapéutico y nutricional. 1st ed. Madrid: Editorial Dilema; 2008.
- [Background] Luabeya KK, Mpontshane N, Mackay M, Ward H, Elson I, Chhagan M, Tomkins A, Van den Broeck J, Bennish ML. Zinc or multiple micronutrient supplementation to reduce diarrhea and respiratory disease in South African children: a randomized controlled trial. PLoS One. 2007 Jun 27;2(6):e541. doi: 10.1371/journal.pone.0000541. PMID 17593956
- [Background] McNair F, Heuchert JWP. Manual for the profile of mood states. San Diego (CA): Educational and Industrical Testing Service; 1971.
- [Background] Mills S, Bone K. The essential guide to herbal safety. 1st ed. Philadelphia: Elsevier; 2005.
- [Background] Maggini S, Wintergerst ES, Beveridge S, Hornig DH. Selected vitamins and trace elements support immune function by strengthening epithelial barriers and cellular and humoral immune responses. Br J Nutr. 2007 Oct;98 Suppl 1:S29-35. doi: 10.1017/S0007114507832971. PMID 17922955